CLINICAL TRIAL: NCT00426335
Title: An Evaluation of a Group CBT Programme for Women With Primary Breast Cancer.
Brief Title: Evaluation of Group CBT Programme With Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Other Study IDs: CCR2839
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Breast Cancer
Keywords: breast; cancer; cognitive behaviour therapy; psychological
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The purpose of this study is to examine whether a group CBT intervention is effective in reducing psychological distress in women with primary breast cancer.

DETAILED DESCRIPTION:
The diagnosis and treatment of cancer is associated with high levels of psychological distress, which can be long-term in duration. The end of adjuvant therapy can be a time which patients find anxiety provoking; as concerns of recurrence and how to return to life after treatment often arise at this juncture.

Cognitive behaviour therapy has demonstrated efficacy in reducing anxiety and depression in people with cancer on a 1:1 basis. The CBT model has been shown to be significantly more beneficial than supportive counselling. Therapy delivered in groups is considered desirable because of its cost effectiveness, and its potential to confer additional benefits in terms of peer support, reduced isolation and modelling of adaptive strategies by other group members.

No studies have looked at the changes in participants health beliefs and beliefs about their ability to copy (self-efficacy) with stress and tolerance of uncertainty following group CBT and the relationship with psychological distress.

The aim of this study is to evaluate a GCBT programme intervention against a waiting list control and to examine its effects on health beliefs, self-efficacy, coping, tolerance of uncertainty and psychological distress in women with early diagnosed breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Primary breast cancer
* post adjuvant treatment

Exclusion Criteria:

* Women with metastatic disease
* Severe cognitive impairment (will not be able to obtain consent or participant in group intervention)
* Inability to complete a questionnaire

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 78 participants in total including 39 female RMH patients with primary breast cancer and are post adjuvant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Estimated)
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Watson, Dr, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden NHS Foundation Trust, London, United Kingdom